CLINICAL TRIAL: NCT07227831
Title: A Phase 2 Study of TheraBionic P1 Device for Patients With Metastatic Hormone Positive Breast Cancer Post Endocrine Therapy
Brief Title: A Ph II Study of the TheraBionic P1 Device in Subjects With Hormone Positive Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Hadeel Assad, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-043
Record Dates: First submitted 2025-11-05; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: HER2-negative Breast Cancer; Hormone Receptor Positive Tumor; Advanced Breast Cancer; Metastatic Breast Cancer
Keywords: therabionic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TheraBionic P1 device (Experimental): Self administered Amplitude-modulated electromagnetic fields three times daily
  Interventions: Device: TheraBionic P1

INTERVENTIONS:
Device: TheraBionic P1 — Amplitude-modulated electromagnetic fields will be self-administered and given continuously to patients in three 60-minute treatments per day, administered in the morning, middle of the day, and in the evening

SUMMARY:
The goal of this clinical trial is to learn if the TheraBionic P1 device given to patients with advanced or metastatic HR positive, HER2 negative breast cancer who have progressed on standard of care options can affect patients survival. The main questions it aims to answer are:

* will the TheraBionic P1 device affect progression free and overall survival in advanced or metastatic HR positive, HER2 negative breast cancer
* the long term safety and tolerability of the TheraBionic P1 device
* assessment of how the disease responded to the TheraBionic P1 device

ELIGIBILITY:
Inclusion Criteria:

* Participant must have locally advanced/unresectable or metastatic Hormone Receptor (HR) positive, Human Epidermal growth factor receptor 2 (HER2) negative breast cancer as defined by the 2010 American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines (estrogen receptor [ER] and/or progesterone receptor [PR] >1% and HER2 negative by immunohistochemistry [IHC] and/or fluorescent in situ hybridization [FISH]).
* Participant must have received and progressed on or are intolerant to all therapies known to confer overall survival benefit, including at least one line of endocrine + CDK4/6 inhibitor therapy AND one line of cytotoxic such as chemotherapy and/or antibody drug conjugates (ADCs).
* Participant must be a woman ≥ 22 years old and must be able to understand and sign an informed consent form.
* Participant must have a life expectancy of at least 3 months.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
* it is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, women of childbearing potential must agree to avoid becoming pregnant starting at initiation of treatment up until at least 30 days after the last TheraBionic P1 session.
* Participants must meet one of the following:

  * Surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy)
  * Post-menopausal, defined as no menses for at least 12 months prior to the screening visit without alternative medical causation.
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence methods such as calendar, ovulation, symptothermal, or post ovulation tracking are not acceptable.
  * Not in a sexual relationship in which they may become pregnant (i.e. same-sex relationship)
  * If they are of childbearing potential, agree to use at least one method of contraception. Withdrawal is not an acceptable contraceptive method.

Exclusion Criteria:

* Participants with known active secondary malignancy, unless, in the opinion of the investigator, it is unlikely to interfere with the safety and efficacy of the endpoints
* Participants that are taking any other investigational drugs.
* Participants that are pregnant or breastfeeding. If a breastfeeding participant would like to be part of this study, breastfeeding must be discontinued.
* Participants with active oral mucosal inflammation, ulceration, or other pathology that could interfere with the use of TheraBionic P1 device (for example: mucositis, thrush, bleeding mucosal lesions, oral herpes, aphthous stomatitis, mouth ulcers, chancre sores, gingivostomatitis, herpangina, aphthae).
* Participants receiving calcium channel blockers and any agent blocking L-type or T-type voltage gated calcium channels (for example: amlodipine, nifedipine, ethosuximide, ascorbic acid/vitamin C, etc.) unless their medical treatment is discontinued at least one day prior to treatment. Participant must agree to abstain from using calcium channel blockers for the duration of treatment on study.
* Participants that do not agree to be followed according to the study protocol or have cognitive or physical inability to use the device.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05-22 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From start of treatment to 5 years after treatment discontinuation or death, whichever comes first
  PFS is defined as the time duration in days from treatment start to progression per physician discretion or death from any cause. Progression will be assessed every 2-3 months for 5 years

SECONDARY OUTCOMES:
Tolerability of the TheraBionic P1 device | From first device use through end of treatment (up to 12 months)
  Tolerability will be assessed by the proportion of participants rated as "tolerating treatment" (yes/no) throughout therapy, based on investigator assessment at each 4-week visit. Participants who discontinue treatment due to device-related symptoms or adverse events will be classified as not tolerating treatment.
Overall Survival (OS) | From start of treatment to 5 years after treatment discontinuation or death, whichever comes first
  The OS is the length of time in days from the start of treatment that participants are still alive and finishing at the date of death from any cause. Participants' survival status will be assessed every 2-3 months for 5 years after the start of TheraBionic P1 treatment.
Overall Response Rate (ORR) | From start of treatment to 5 years after treatment initiation or death, whichever comes first
  The ORR is calculated as the proportion of participants with complete response (CR) or partial response (PR) per physician discretion. ORR will be assessed every 2-3 months for 5 years after the start of TheraBionic P1 treatment.
Disease control rate (DCR) | From start of treatment to 5 years after treatment initiation or death, whichever comes first
  DCR is defined as the proportion of participants with complete response (CR), partial response (PR), or stable disease (SD) per physician discretion. DCR will be assessed every 2-3 months for 5 years after the start of TheraBionic P1 treatment.
Duration of response (DOR) | From start of treatment to 5 years after treatment initiation or death, whichever comes first
  DOR will be measured as the amount of time from the time of response until the first date of progressive disease (PD) per physician discretion. Participants' progression status will be assessed every 2-3 months for 5 years after the start of TheraBionic P1 treatment.
Time to progression (TTP) | From start of treatment to 5 years after treatment initiation or death, whichever comes first
  Time to progression will be recorded in days starting from TheraBionic P1 treatment initiation and finishing at the date of progression per physician discretion.

IPD SHARING:
Plan to Share IPD: Undecided